CLINICAL TRIAL: NCT06914193
Title: Intravenous Infusion of Esketamine in Combination With Pulsed Radiofrequency of Dorsal Root Ganglion for Postherpetic Neuralgia
Brief Title: Esketamine Combined With PRF of DRG for Postherpetic Neuralgia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Xiaotangshan Hospital (Other); The First Hospital of Fangshan District,Beijing (Other); Beijing Ditan Hospital (Other); Hengshui People's Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Day surgery and Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY-2024-332-02-05
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Postherpetic Neuralgia
Keywords: Postherpetic Neuralgia; Esketamine
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- esketamine group (Experimental): esketamine+PRF group
  Interventions: Drug: esketamine+PRF treatment group
- control group (Active Comparator): PRF group
  Interventions: Drug: PRF treatment group

INTERVENTIONS:
Drug: esketamine+PRF treatment group — In the esketamine group, in addition to receiving PRF treatment+pregabalin, patients will also undergo a single intravenous infusion of esketamine.
  Other Names: esketamine+PRF treatment+pregabalin
  Arms: esketamine group
Drug: PRF treatment group — In the control group, patients will receive PRF treatment. PRF will be performed on DRG by an designated physician in each participating center. The patients will be treated with PRF (PMG-230, Baylis Medical Inc.) using a 21-gauge sterilized radiofrequency needle (a 10-cm trocar with a 5-mm active tip, PMF-21-100-5, Baylis Medical Inc.), which will be carefully inserted until the needle tip reached the upper edge of the intervertebral foramen under the guidance of three-dimensional (3D) CT. PRF treatment (PMG-230, Baylis Medical Inc.) targeting to DRG will be applied for 900 seconds. The parameters of PRF treatment will be set at 42 ℃, 2 Hz with 20 milliseconds current. Regarding pregabalin, the dosage is titrated based on patients'pain intensity and tolerance. This process fully accounts for individual patient differences to optimize treatment outcomes.
  Other Names: PRF treatment+pregabalin
  Arms: control group

SUMMARY:
This trial's primary objective is to compare the analgesic efficacy of esketamine in combination with pulsed radiofrequency (PRF) of dorsal root ganglion(DRG) against that of PRF monotherapy in patients with postherpetic neuralgia(PHN).

DETAILED DESCRIPTION:
This study aims to determine whether the addition of esketamine to the PRF of DRG regimen can relieve pain in PHN patients. By doing so, the research endeavors to identify a rapid, effective, and safe treatment approach for refractory PHN patients

ELIGIBILITY:
Inclusion Criteria:

1. Ages more than 18 years;
2. Pain persisting for over three months following the onset of the herpes zoster skin rash;
3. Lesions located in in the unilateral cervical, thoracic, and lumbosacral segments;
4. Having an average pain score of at least 4 on a Numeric Rating Scale (NRS, 0 = no pain, 10= worst possible pain)； Planned to perform CT-guided PRF treatment of the Dorsal root ganglion（DRG）

Exclusion Criteria:

1. Obstructive sleep apnoea syndrome;
2. Those who receive other more invasive treatments, such as radiofrequency thermocoagulation (RFT) of DRG.
3. A history of systemic immune diseases, organ transplantation, or cancers;
4. A history of severe cardiopulmonary, hepatic, renal dysfunction or coagulation function disorder;
5. A history of schizophrenia, epilepsy, or myasthenia gravis, delirium;
6. Comorbid hyperthyroidism or phaeochromocytoma;
7. Recent history of drug abuse;
8. Having contraindications to esketamine;
9. Communication difficulties.
10. Women who are preparing for pregnancy, in the pregnancy or lactation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
The primary comparison is the difference between the means of the daily mean pain scores over the first 7 days, measured on an 11-point NRS | 7-day period
  The Numeric Rating Scale (NRS) score is a way to quantify the degree of subjective feelings such as pain using numbers. Generally, 0 represents no pain, and 10 represents the most severe pain.A higher score indicates more severe pain

SECONDARY OUTCOMES:
average weekly NRS score | up to 12 weeks
  Generally, 0 represents no pain, and 10 represents the most severe pain.A higher score indicates more severe pain
Averaged weekly analgesic consumption | up to 12 weeks
  Averaged weekly consumption per analgesic of each participant for rescue analgesia
the 12-item Short-Form Health Survey (SF-12) score | At the end of weeks1, 2, 4, 8, and 12 after treatment
  Quality of life (QoL) assessed by the SF-12 score (range 0-100, with higher scores indicating better health status)
the Pittsburgh Sleep Quality Index (PSQI) score | At the end of weeks 1,2, 4, 8, and 12 after treatment
  Sleep quality measured by PSQI score (range 0-21, with higher scores indicating poorer sleep quality).
the Patient Global Impression of Change scale (PGIC) | At the end of weeks 1,2 4, 8, and 12 after treatment
  The proportion of patients with a response of "no change", "minimally improved", "much improved" or "very much improved" on PGIC.
The Hospital Anxiety and Depression Scale (HADS) | At the end of weeks 1, 2, 4, 8, and 12 after treatment
  It consists of two sub-scales. Each sub-scale consists of 7 items and each item scored from 0 to 3. A higher score indicates more severe anxiety or depression. A score of 11 or above can indicate clinically significant anxiety or depression.
Safety assessments | Conducted on Day 0, Day 1, Day 3, and at the end of weeks 1, 2, 4, 8, and 12 after treatment
  intraoperative complications, PRF-related complications, Eskatamine-related complications, Pregabaline-related complications
success rate | At the end of weeks 1, 2, 4, 8, and 12 after treatment
  The success rate is defined as more than a 50% reduction in NRS-11 score.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Not yet decided